CLINICAL TRIAL: NCT03353116
Title: The Assessment of Maxillary Stability in Bimaxillary Orthognathic Patients Treated by Mandible-first Approach Versus Maxilla-first Approach; Randomized Controlled Clinical Trial
Brief Title: Assessment of Maxillary Stability in Bimaxillary Orthognathic Patients Using the Inverted Sequence Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Hamdy, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2017-11-16
Record Dates: First submitted 2017-11-09; First posted 2017-11-27 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Class III Malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class III

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- maxilla first group (Active Comparator): the maxillary osteotomy is going to be done and fixed first
  Interventions: Procedure: the maxilla first
- mandible first group (Experimental): the mandibular osteotomy is going to be done and fixed first
  Interventions: Procedure: the mandible first

INTERVENTIONS:
Procedure: the mandible first — the mandible osteotomy is going to be done and fixed first
  Other Names: the inverted sequence
  Arms: mandible first group
Procedure: the maxilla first — the maxilla osteotomy is going to be done and fixed first
  Other Names: the regular sequence
  Arms: maxilla first group

SUMMARY:
The investigator will assess the inverted sequence approach in the treatment of class III patient undergoing bimaxillary orthognathic surgery

DETAILED DESCRIPTION:
The investigator will compare the maxillary stability in class III orthognathic patients undergoing bimaxillary surgery by two surgical approaches ; the mandible-first (intervention) and the maxilla-first (control)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with skeletal class III malocclusion requiring bimaxillary orthognathic surgery
2. Patients free from any systemic disease
3. Patients who approved to be included in the trial and signed the informed consent
4. Patients with no signs or symptoms of temporomandibular disorders.

Exclusion Criteria:

1. Patients with cleft lip and palate "can have an unfavorable effect on facial growth (LARRY M. WOLFORD, 2002)"
2. Patients receiving chemotherapy or radiotherapy "due to the risk of low bone quality and healing (JW, 2003) "
3. Patients who refused to be included in the trial

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
the change in maxilla stability | 6 months
  to assess the change in maxillary stability on cone beam CT obtained immediately and 6 month postoperative.
  the measuring unit is millimeter

SECONDARY OUTCOMES:
Patient satisfaction | 6 month
  "the quality of life questionnaire" describes the patient's satisfaction during the entire treatment period which is done through a questionnaire answered by the patient through a score between 0-10 the measuring unit is numerical

CONTACTS AND LOCATIONS:
Overall Officials: mohamed mh hamdy, master, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Middle East, Egypt

IPD SHARING:
Plan to Share IPD: No
after the completion of my research i will publish the data in an international journal

REFERENCES:
- [Background] Esteves LS, Castro V, Prado R, de Moraes e Silva CA, do Prado CJ, Trindade Neto AI. Assessment of skeletal stability after counterclockwise rotation of the maxillomandibular complex in patients with long-face pattern subjected to orthognathic surgery. J Craniofac Surg. 2014 Mar;25(2):432-6. doi: 10.1097/SCS.0000000000000395. PMID 24531245
- [Background] Ann HR, Jung YS, Lee KJ, Baik HS. Evaluation of stability after pre-orthodontic orthognathic surgery using cone-beam computed tomography: A comparison with conventional treatment. Korean J Orthod. 2016 Sep;46(5):301-9. doi: 10.4041/kjod.2016.46.5.301. Epub 2016 Sep 19. PMID 27668193
- [Background] Beziat JL, Babic B, Ferreira S, Gleizal A. [Justification for the mandibular-maxillary order in bimaxillary osteotomy]. Rev Stomatol Chir Maxillofac. 2009 Dec;110(6):323-6. doi: 10.1016/j.stomax.2009.09.009. Epub 2009 Nov 25. French. PMID 19939425
- [Background] Liebregts J, Baan F, de Koning M, Ongkosuwito E, Berge S, Maal T, Xi T. Achievability of 3D planned bimaxillary osteotomies: maxilla-first versus mandible-first surgery. Sci Rep. 2017 Aug 24;7(1):9314. doi: 10.1038/s41598-017-09488-4. PMID 28839184

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-23): https://cdn.clinicaltrials.gov/large-docs/16/NCT03353116/Prot_SAP_001.pdf
  • Informed Consent Form (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/16/NCT03353116/ICF_000.pdf